CLINICAL TRIAL: NCT05750927
Title: Aortic Stenosis With COmplex PCI (ASCOP) Features Retrospective Registry on Contemporary Management and Outcomes
Acronym: ASCOP
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 723-1412202
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement; Angioplasty, Balloon, Coronary; Coronary Artery Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease | interventions — Transcatheter Aortic Valve Replacement; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASCoP (severe Aortic Stenosis with Complex PCI features): Subjects with severe aortic stenosis undergoing transcatheter aortic valve intervention and with concomitant, complex coronary artery disease with a clinical indication for percutaneous coronary intervention
  Interventions: Procedure: Transcatheter aortic valve intervention (TAVI) and percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Transcatheter aortic valve intervention (TAVI) and percutaneous coronary intervention (PCI) — TAVI and PCI to be administered as per physician's indication and choice, in one or more stages

SUMMARY:
To describe the prevalence and clinical features of patients with severe aortic stenosis undergoing TAVI and concomitant clinically indicated, complex and/or high-risk PCI

DETAILED DESCRIPTION:
The aims of this study are:

* to describe the prevalence and clinical features of patients with severe aortic stenosis undergoing TAVI and concomitant clinically indicated, complex and/or high-risk PCI
* to depict the different possible strategies that are currently employed in this context and to retrospectively analyze outcomes
* to investigate predictors of better outcomes

ELIGIBILITY:
1. Severe, symptomatic aortic stenosis with an indication to TAVI
2. Concomitant, stable CAD with an indication to complex PCI, as anticipated by angiography, defined as follows (one or more features)

   1. Left-main (LM) CAD or proximal left anterior descending (LAD) / left circumflex (LCx) lesions requiring LM-PCI
   2. Three-vessel disease
   3. Last remaining vessel
   4. Bifurcation PCI (proximal bifurcation)
   5. Severely calcified lesions requiring calcium plaque modification (rotational/orbital atherectomy, intravascular lithotripsy, scoring or cutting balloon)
   6. Lesion length > 30 mm
   7. Severely depressed Left ventricular function requiring mechanical circulatory support (intra-aortic balloon pump - IABP, Impella, Extracorporeal Membrane Oxygenation - ECMO

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe, symptomatic aortic stenosis with an indication to TAVI 2. Concomitant, stable CAD with an indication to complex PCI, as anticipated by angiography, defined as follows (one or more features)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
POCE | 1 year
  all-cause deaths, strokes (any), myocardial infarction and major bleedings

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Montalto C, Munafo AR, Soriano F, Arslani K, Brunner S, Verhemel S, Cozzi O, Mangieri A, Buono A, Squillace M, Nava S, Diez Gil JL, Scotti A, Foroni M, Esposito G, Mandurino-Mirizzi A, Bauer D, Ornelas B, Codner P, Piayda K, Porto I, Marco F, Sievert H, Kornowski R, Tousek P, Fischetti D, Latib A, Sanchez JS, Maffeo D, Bedogni F, Reimers B, Regazzoli D, Mieghem NV, Sondergaard L, Saia F, Toggweiler S, Backer O, Oreglia JA. Outcomes of complex, high-risk percutaneous coronary intervention in patients with severe aortic stenosis: the ASCoP registry. EuroIntervention. 2025 Apr 21;21(8):e426-e436. doi: 10.4244/EIJ-D-24-00933. PMID 40259842